CLINICAL TRIAL: NCT00097903
Title: Phase 1 Trial of Oral Karenitecin® in Patients With Solid Tumors"
Brief Title: Trial of Oral Karenitecin in Patients With Solid Tumors and Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioNumerik Pharmaceuticals, Inc. (Industry)
Collaborators: Crown Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: KTN22208
Record Dates: First submitted 2004-12-01; First posted 2004-12-02 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Carcinoma; Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; Solid Tumors; Oral
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — cositecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Karenitecin IV/ Karenitecin tablet
  Interventions: Drug: Karenitecin (BNP1350)

INTERVENTIONS:
Drug: Karenitecin (BNP1350) — Phase 1 study,dose-escalation design
  Other Names: Karenitecin also referred to as BNP1350

SUMMARY:
The purpose of this study is to determine the maximum safe dose of orally administered Karenitecin (BNP1350) in patients with solid tumors.

DETAILED DESCRIPTION:
Initially, the safety, side effects and recommended phase 2 dose of oral Karenitecin in patients with advanced solid tumors will be determined.

When the recommended phase 2 dose has been determined, the specified dose will be used to determine if Karenitecin is effective in the treatment of patients with relapsed or refractory non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria

* Patients entering the Phase 1 portion of the study must have a histologically or cytologically documented diagnosis of cancer (solid tumors) refractory to conventional therapeutic modalities or for which no conventional treatment exists.
* Patients entering the Phase 2 portion of the study must have a histologically or cytologically documented diagnosis of advanced (Stage IIIb/IV) NSCLC.
* Patients entering the Phase 1 portion of the study can have either measurable or evaluable disease.
* Patients entering the Phase 2 portion of the study must have measurable disease meeting RECIST criteria.
* Patients must have an ECOG performance status of less than or equal to 1.
* More than 2 weeks must have elapsed since previous chemotherapy and 6 weeks from previous treatment with nitrosoureas or mitomycin-C.
* Patients must have fully recovered from the toxic effects of prior therapy.
* Patients entering the Phase 1 portion of the study may have received up to two prior chemotherapy programs including adjuvant or neoadjuvant therapy.
* Patients entering the Phase 2 portion of the study may have received only one prior chemotherapy program including adjuvant or neoadjuvant therapy for NSCLC.
* More than 2 weeks must have elapsed since previous radiation therapy and prior radiation must be less than or equal to 15% of the bone marrow.
* Required Initial Laboratory Data: *ANC ≥ 1,500/mm3, *Platelet count ≥ 100,000/mm3, *SGPT < 1.5 times ULN, *Alkaline phosphatase < 2.0 times ULN, *Bilirubin < 1.5 mg/dl, *Serum creatinine < 1.5 times ULN

Exclusion Criteria:

* Pregnant or lactating women.
* Uncontrolled high blood pressure, uncontrolled diabetes mellitus, unstable angina, symptomatic congestive heart failure (CHF), myocardial infarction (MI) within 6 months, or uncontrolled arrhythmia.
* Phase 2 no previous or concurrent malignancy
* Central Nervous System (CNS) metastasis if neurologically unstable or requiring steroid use.
* Active infection.
* Known positive HIV status.
* Conditions requiring use of H2 blockers or other antacids.
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-05; Primary Completion 2011-10 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Overall Safety and determination of MTD, and recommended Phase 2 dose | throughout study

SECONDARY OUTCOMES:
Pharmacokinetics | various timepoints
Tumor response | various timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- Ellis Fischel Cancer Center, Columbia, Missouri, United States